CLINICAL TRIAL: NCT04526379
Title: Communication in Prader-Willi Syndrome: Study of Emotional Control Related to Behavioral Disorders, Their Daily Repercussions and Examination of an Innovative Therapy: Transcutaneous Electrical Nerve Stimulation of the Vagus Nerve - PRACOM1
Brief Title: Study of Emotion and Cognition Abilities of Children With PWS and Proposition of an Innovative Remediation
Acronym: PRACOM1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/18/0335
Record Dates: First submitted 2020-03-03; First posted 2020-08-25 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Prader-Willi Syndrome
Keywords: Emotion; Cognition
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: The study consists of 2 parts. The first part compares 30 children with PWS compared to 30 control children without PWS. The second part will be based on 12 children with PWS who have undergone part 1.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- children with PWS (Experimental): Evaluation of cognitive abilities of children with PWS by several cognitive tasks and neuropsychological tests.
  Interventions: Behavioral: Questionnaires; Device: t-VNS
- non affected children (Other): Evaluation of cognitive abilities of children with PWS compared to a non-pathologic population of children by several cognitive tasks and neuropsychological tests
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Evaluation of behavioral disorders of children with PWS by questionnaires
Device: t-VNS — Evaluation of the influence of 6 month-stimulation by t-VNS on emotional, cognitive, and behavioral/clinical characteristics of 12 children with PWS on 30 PWS patients included.
  Arms: children with PWS

SUMMARY:
The present project project is divided in two parts. The primary aim of the part 1 of this study is to evaluate emotional control abilities of children with Prader-Willi syndrome (PWS) aged from 9 to 15 years and to study repercussions of this supposed lack of abilities on cognitive capacities and behavioral troubles. The study also evaluate influence of the emotional symptomatology of patients on quality of parents' life and on the care of parents and scholar/institutional caregivers. In the second part of this study, the study evaluate the feasibility and the tolerance to a non-invasive device supposed to reduce emotional symptoms in this disease.

DETAILED DESCRIPTION:
Prader-Willi Syndrome (PWS) is a rare genetic disorder involving a variety of clinical, behavioral and cognitive symptoms. 83 to 97% of patients have episodes of temper tantrum, associated with an important emotional lability. These different cognitive and behavioral limitations are barriers to the social integration of patients. The PWS also has repercussions on well-being and quality of life of the family. Thus, the present project focuses on the characteristics of emotional control related to the anger of children with PWS and its behavioral, cognitive and social implications. In addition, at a therapeutic level, our project assumes that transcutaneous electrical nerve stimulation (t-VNS), a non-invasive, safe and inexpensive method, could be effective in reducing the severity of behavioral disorders such as temper tantrums while improving cognitive performance and social communication in the PWS.

ELIGIBILITY:
Inclusion Criteria:

* Age from 9 to 15 years old
* Prader-Willi syndrome with identified genotype.
* No psychiatric disorder neither PWS.
* Severe global symptomatology attested by a CGI-S score

Exclusion Criteria:

* Identified psychiatric or behavioral disorders
* Severe visual or hearing impairment.
* Sleep apnea syndrome treated with non-invasive ventilation,
* Epileptic seizures
* Cardiac disorders.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
assessment of the level of emotional control | day 0
  composite score of emotional control level of children with PWS composed of scores of emotional lability

SECONDARY OUTCOMES:
Evaluation of behavioral disorders of children with PWS by CBCL (Child Behavior Checklist) scale | month 6
  CBCL (Child Behavior CheckList) scale: is a questionnaire comprising 1) an adaptive functioning scale (activities, social and school spheres), 2) a syndrome scale (social withdrawal, anxiety / depression, somatic complaints, social problems, thinking problems, attention problems, behavior problems and aggressiveness; total of internalized problems and total of externalized problems), 3) a DSM-oriented scale (Lengua et al., 2001; anxiety, attention problems / hyperactivity, behavior problems, depression, opposition / mistrust, social problems / immaturity, somatization). (duration = 20 ') - there is no minimum and maximum values as this is an evaluation of behavioral disorders
Evaluation of behavioral disorders of children with PWS by Hyperphagia Questionnaire | month 6
  HQ-CT (Hyperphagia Questionnaire) scale: The HQ-CT (Hyperphagia Questionnaire for Use in Prader-Willi Syndrome Clinical Trials, Fehnel et al., 2015, appendix 10) is a scale derived from the Dykens hyperphagia questionnaire (Dykens et al., 2007). The specificity of the Dykens questionnaire makes it a favored tool in the international literature in the evaluation of the eating behavior of patients with PWS (Crain, 2010). The HQ-CT was created specifically to assess the eating behavior of these patients in clinical trials. It consists of 9 items for which a person taking care of the patient (family or caregiver) indicates the frequency and severity of the behavior described on a 5-point Likert scale (with 1 = absence of the behavior and 5 = very frequent behavior or severe) (⍺ = .91). (duration = 5 ') - so 1 is the minimum value and 5 the maximum value and higher scores mean a worse outcome
Evaluation of cognitive abilities of children with PWS | 2 days
  emotional language task
Test of evaluation of cognitive abilities | 2 days
  multimodal emotional recognition test MERT
Evaluation of cognitive abilities | 2 days
  WISC-V

CONTACTS AND LOCATIONS:
Overall Officials: Maithé TAUBER, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, France